CLINICAL TRIAL: NCT01656551
Title: A Factorial Study Comparing Pemetrexed With Gemcitabine and Testing the Efficacy of the Addition of Cisplatin in Elderly Patients With Non Squamous Advanced, Metastatic or Recurrent NSCLC.
Brief Title: MILES-4: Study Comparing Gemcitabine and Pemetrexed, With or Without Cisplatin, in Patients With Nonsquamous Lung Cancer
Acronym: MILES-4
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Cancer Institute, Naples (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: MILES-4; 2012-000164-25 (EudraCT Number)
Record Dates: First submitted 2012-07-23; First posted 2012-08-03 (Estimated); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Non-small Cell Lung Cancer Metastatic; Non-small Cell Lung Cancer Stage IIIB
Keywords: elderly; chemotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Gemcitabine; Pemetrexed; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- A: Gemcitabine (Active Comparator): Single agent gemcitabine dose 1200 mg/m2 days 1 and 8, every 3 weeks
  Interventions: Drug: Gemcitabine
- B: Gemcitabine + Cisplatin (Experimental): Gemcitabine dose 1000 mg/m2 days 1 and 8, every 3 weeks
  Interventions: Drug: Gemcitabine; Drug: Cisplatin
- C: Pemetrexed (Active Comparator)
  Interventions: Drug: Pemetrexed
- D: Pemetrexed + Cisplatin (Experimental)
  Interventions: Drug: Pemetrexed; Drug: Cisplatin

INTERVENTIONS:
Drug: Gemcitabine
  Arms: A: Gemcitabine; B: Gemcitabine + Cisplatin
Drug: Pemetrexed — 500 mg/m2 day 1 every 3 weeks
  Arms: C: Pemetrexed; D: Pemetrexed + Cisplatin
Drug: Cisplatin — 60 mg/m2 day 1 every 3 weeks
  Arms: B: Gemcitabine + Cisplatin; D: Pemetrexed + Cisplatin

SUMMARY:
The purposes of this study are to test whether the addition of cisplatin to single agent chemotherapy (either gemcitabine or pemetrexed) prolongs survival in elderly patients with non squamous non small cell lung cancer (NSCLC), and to test whether pemetrexed prolongs survival as compared to gemcitabine in elderly patients with non squamous NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cytologically or histologically confirmed non-small cell lung cancer.
* Non squamous tumor type (including those with a non-specified tumor type).
* Metastatic (stage IV, both M1A or M1B) or locally advanced (stage IIIB, with metastasis to supraclavicular nodes) according to TNM VII edition.
* Both patients at first diagnosis or those with disease recurrence after former surgery are eligible.
* At least one target or non-target lesion according to RECIST revised version 1.1.
* Male or female > or = 70 years of age.
* ECOG PS 0 or 1.
* Life expectancy > 3 months.
* Neutrophils > or = 1500 mm3, platelets > or = 100000 mm3, and haemoglobin > or = 9 g/dL.
* Bilirubin level either normal or < 1.5 x ULN.
* AST (SGOT) and ALT (SGPT) < or = 2.5 x ULN (< or = 5 x ULN if liver metastasis are present).
* Serum creatinine < 1.5 x ULN.
* Signed written informed consent.

Exclusion Criteria:

* Prior chemotherapy or therapy with systemic anti-neoplastic therapy for advanced disease. Prior surgery and/or localised irradiation is permitted. Prior adjuvant chemotherapy is permitted if it did not contain gemcitabine and pemetrexed and if at least 6 months elapsed from the end of adjuvant chemotherapy.
* Any unstable systemic disease (including active infections, significant cardiovascular disease or myocardial infarction within the previous year, any significant hepatic, renal or metabolic disease), metabolic dysfunction, physical examination finding, or clinical laboratory finding that contraindicates the use of study medications or render the patient at high risk from treatment complications.
* Any other malignancies within 5 years (except for adequately treated carcinoma in situ of the cervix or basal or squamous cell skin cancer or surgically resected prostate cancer with normal PSA).
* Patients with symptomatic brain metastasis or spinal cord compression that has not yet been treated with surgery and/or radiation; patients with CNS metastases or spinal cord compression previously treated with surgery and/or radiation are eligible if they are asymptomatic and do not require steroids (anti-seizure medications are allowed).
* Known or suspected hypersensitivity to any of the study drugs

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 232 (Actual)
Dates: Start 2012-08 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
overall survival | one year
  factorial design with two comparisons: single agent chemotherapy versus chemotherapy plus cisplatin (Arms A+C versus Arms B + D), and gemcitabine versus pemetrexed (Arms A+B versus Arms C+D)

SECONDARY OUTCOMES:
worst grade toxicity per patient | evaluated at end of each 3 week cycle of chemotherapy up to 18 weeks
  according to Common Toxicity Criteria for Adverse Events v. 4.03
progression free survival | 6 months
changes in quality of life | baseline and up to 18 weeks
objective response | after 9 and 18 weeks of therapy

OTHER OUTCOMES:
identification of patient and lesion specific prognostic factors | 2 years
identification of patient and lesion specific factors predictive of chemotherapy efficacy | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Cesare Gridelli, M.D., Principal Investigator — S.G. Moscati Hopital, Avellino, Italy, Division of Medical Oncology; Francesco Perrone, M.D., Ph.D, Principal Investigator — National Cancer Institute Naples, Italy; Director Clinical Trials Unit; Ciro Gallo, M.D., Ph.D, Principal Investigator — Second University of Naples, Italy; Chair of Medical Statistics; Massimo Di Maio, M.D., Principal Investigator — National Cancer Institute, Naples
Locations (48):
- Italy (48):
  - Ospedale San Lazzaro, Alba
  - Ospedali Riunit Umberto I-Lancisi-Salesi, Ancona
  - Oncologia Universitaria degli Studi di Roma, Aprilia
  - Ospedale Cardinal Massaia, Asti
  - S. Giuseppe Moscati, Avellino
  - Ospedale Senatore Antonio Perrino, Brindisi
  - Univeristaria Policlinico Monserrato di Cagliari, Cagliari
  - Ospedale A. cardarelli, Campobasso
  - U.L.S.S. 15 Veneto, Camposampiero
  - Ospedale Ramazzini di Carpi, Carpi
  - Azienda Ospedaliera Garibalda Nesimadi Catania, Catania
  - Policlinico vittorio Emanuele, Catania
  - Ospedale della Madonna della Navicella, Chioggia
  - Ospedale Civile di Faenza, Faenza
  - Ospedale Fabrizio Spaziani, Frosinone
  - IRCCS AOU San Martino IST Genova, Genova
  - Ospedale Villa Scassi, Genova
  - Azienda Ospedaliera Vito Fazzi, Lecce
  - Ospedale Civile di Legnano, Legnano
  - Ospedale Umberto I, Lugo
  - IRCCS-Meldola, Meldola
  - Ospedale L. Sacco Polo Universitario, Milan
  - Ospedale S. Paolo, Milan
  - U.L.S.S. 13, Mirano
  - H San Gerardo, Monza
  - A.O.U. Federico II, Napoli
  - Istituto Nazionale dei Tumori, Napoli
  - Ospedale Cardirelli, Napoli
  - Seconda Università di Napoli, Napoli
  - Istituto Sacro Cuore Don Calabria, Negrar
  - Istituto Oncologico Veneto, Padua
  - Ospedale Civile Umberto I, Pagani
  - Azienda Ospedaleira Ospedali Riuniti Villa Sofia Cervello, Palermo
  - Casa di cura La Maddalena, Palermo
  - Fondazione Salvatore Maugeri, Pavia
  - A.O. San Carlo, Potenza
  - Irccs - Crob, Rionero in Vulture
  - AO San Camillo Forlanini, Roma
  - Campus Biomedico, Roma
  - Ospedale S. Giovanni Calibita Fatebenfratelli, Roma
  - Ospedale Guglielmo da Saliceto-USL di Piacenza, Saliceto
  - Oncologia IRCCS - Casa Sollievo Sofferenza, San Giovanni Rotondo
  - A.O. di Busto Arsizio, Saronno
  - Ospedale di Sondrio, Sondrio
  - Ospedale SS. Trinità, Sora
  - Ospedale S. Andrea, Vercelli
  - Ospedale S. Bortolo, Vicenza
  - ASL Viterbo Ospedale Belcolle, Viterbo

REFERENCES:
- [Derived] Gridelli C, Morabito A, Cavanna L, Luciani A, Maione P, Bonanno L, Filipazzi V, Leo S, Cinieri S, Ciardiello F, Burgio MA, Bilancia D, Cortinovis D, Rosetti F, Bianco R, Gebbia V, Artioli F, Bordonaro R, Fregoni V, Mencoboni M, Nelli F, Riccardi F, di Isernia G, Costanzo R, Rocco G, Daniele G, Signoriello S, Piccirillo MC, Gallo C, Perrone F. Cisplatin-Based First-Line Treatment of Elderly Patients With Advanced Non-Small-Cell Lung Cancer: Joint Analysis of MILES-3 and MILES-4 Phase III Trials. J Clin Oncol. 2018 Sep 1;36(25):2585-2592. doi: 10.1200/JCO.2017.76.8390. Epub 2018 Jul 20. PMID 30028656